CLINICAL TRIAL: NCT05176678
Title: Clinical Proof-of-concept Study on Immunological Effects of Consuming Increasing Doses of a Natural Peptide in Healthy Volunteers
Brief Title: Immunological Effect of Increasing Doses of Natural Peptide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research Director, Natural Immune Systems Inc
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: NIS 184-001
Record Dates: First submitted 2021-11-04; First posted 2022-01-04 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escalating dose of natural protein hydrolysate - sequence A (Active Comparator): Participants will consume escalating doses of natural protein hydrolysate: Week 1-2: 1 gram/day, Week 3-4: 2 gram/day, Week 5-6: 4 gram/day.
  Interventions: Dietary Supplement: 1 gram of a protein hydrolysate; Dietary Supplement: 2 grams of a protein hydrolysate; Dietary Supplement: 4 grams of a protein hydrolysate
- Escalating dose of natural protein hydrolysate - sequence B (Active Comparator): Participants will consume escalating doses of natural protein hydrolysate: Week 1-2: 1 gram/day, Week 3-4: 2 gram/day, Week 5-6: 8 gram/day.
  Interventions: Dietary Supplement: 1 gram of a protein hydrolysate; Dietary Supplement: 2 grams of a protein hydrolysate; Dietary Supplement: 8 grams of a protein hydrolysate

INTERVENTIONS:
Dietary Supplement: 1 gram of a protein hydrolysate — After 1 gram of a protein hydrolysate is taken daily for 2 weeks, 1 blood draw will be taken.
Dietary Supplement: 2 grams of a protein hydrolysate — After 2 grams of a protein hydrolysate is taken daily for 2 weeks, 1 blood draw will be taken.
Dietary Supplement: 4 grams of a protein hydrolysate — After 4 grams of a protein hydrolysate is taken daily for 2 weeks, 1 blood draw will be taken.
  Arms: Escalating dose of natural protein hydrolysate - sequence A
Dietary Supplement: 8 grams of a protein hydrolysate — After 8 grams of a protein hydrolysate is taken daily for 2 weeks, 1 blood draw will be taken.
  Arms: Escalating dose of natural protein hydrolysate - sequence B

SUMMARY:
A trial monitoring the immune effects in 24 people with 4 different doses (1 gram per day, 2 grams per day, 4 grams per day, 8 grams per day) of a natural plant-based protein hydrolysate.

DETAILED DESCRIPTION:
The goal for this clinical proof-of-concept study is to compare immune effects of a novel plant-based peptide on IL-17, Th17 and related immunological mechanisms.

An open-label, escalating dose study design monitoring immune effects in which healthy men and women take doses of a natural protein hydrolysate daily for 6 weeks.

During the first 2 weeks, participants will consume 1 gram/day. For the next 2 weeks, participants will consume 2 grams/day. For the final 2 weeks, participants will be randomly assigned to consume either 4 grams/day or 8 grams/day.

Blood samples are collected at baseline and every 2 weeks. The blood will be used for testing of the numbers of T lymphocytes that secrete Interleukin-17 after ex vivo cell cultures.

ELIGIBILITY:
Inclusion Criteria:

* 24 men and women
* Eating a typical diet that does not exceed an estimated average of 9 grams of salt per day;
* Willing to comply with a 24-hour wash-out period for vitamins and nutritional supplements;
* Willing to comply with study procedures including: Maintaining a consistent diet and lifestyle routine throughout the study, Consistent habit of bland breakfasts on days of clinic visits, Abstaining from exercising and nutritional supplements on the morning of a study visit, Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit; Abstaining from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery Vaccination during past month;
* Vaccination planned during study;
* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Diagnosed with an autoimmune disorder;
* Diagnosed with obstructive sleep apnea syndrome (OSAS);
* Currently taking medication containing Levodopa (L-dopa);
* Having received a cortisone shot within the past 6 months;
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/life changes;
* Currently in intensive athletic training (such as marathon runners);
* An unusual sleep routine
* Changes to nutritional supplements during the past month;
* Currently taking Vitamin D at a dose higher than 1,000 IU/day;
* Currently taking omega-3 at a dose higher than 1 gram/day;
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Women of childbearing potential: Pregnant, nursing, or trying to become pregnant;
* Known food intolerances related to ingredients in active test product.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-11-04 (Estimated); Study Completion 2023-07-11 (Estimated)

PRIMARY OUTCOMES:
Changes to ex vivo PHA-mediated Th-17 cytokine secretion | 2 weeks, 4 weeks, 6 weeks
  Ex vivo PBMC cultures with the mitogen PHA, followed by testing of cytokine production using a Th-17 Luminex array.

SECONDARY OUTCOMES:
Evaluation of lymphocytes | 2 weeks, 4 weeks, 6 weeks
  Ex vivo PBMC cultures with the mitogen PHA, followed by flow cytometry evaluation of T-cell differentiation and intracellular staining for Interleukin-17.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte S Jensen, Principal Investigator — NIS Labs
Locations (1):
- Gitte Jensen, Klamath Falls, Oregon, United States